CLINICAL TRIAL: NCT06103526
Title: Immunonutrition and Enhanced Recovery After Surgery Protocols in Gynecologic Oncology
Brief Title: Immunonutrition in ERAS Protocols in Gynecologic Oncology
Acronym: NUTRIGO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Nikolaos Thomakos, Associate Professor of Obstetrics and Gynecology, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1233456
Record Dates: First submitted 2023-10-16; First posted 2023-10-26 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Nutritional Deficiency; Gynecologic Cancer; ERAS
MeSH Terms: conditions — Malnutrition | interventions — Immunonutrition Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunonutrition and ERAS (Active Comparator): Immunonutrition supplements will be provided to patients in the form of oral supplements given twice daily for 3 days pre-surgery and 3 days post-surgery.
  Interventions: Dietary Supplement: Immunonutrition
- ERAS without immunonutrition (No Intervention): Typical ERAS protocol will be followed for patients in that group

INTERVENTIONS:
Dietary Supplement: Immunonutrition — enteral supplementation with high amount of proteins, arginine, glutamine, nonessential fatty acids, branched chain fatty acids, nucleotides, or RNA
  Arms: Immunonutrition and ERAS

SUMMARY:
A patient with oncological pathology of any type because of impaired digestion and nutrient absorption, decreased intake, and increased nutrition requirements has an increased risk of malnutrition and moderate to severe weight loss.In the present study the investigators will evaluate the impact of perioperative immunonutrition supplementation on the postoperative outcomes.

DETAILED DESCRIPTION:
Malnutrition has a major effect not only on the postoperative course of cancer surgery but can also complicate or even limit administration or compromise the effectiveness of other treatments such as chemotherapy or radiotherapy in the perioperative period. Immunonutrition is a type of artificial nutrition based on the use of some types of macro- or micronutrients.The purpose of this review was to evaluate the use, indications, and effects of these formulas in oncologic surgical patients in real time and to identify the types of patients who can benefit from enteral immunonutrition.

ELIGIBILITY:
Inclusion Criteria:

* women with any gynaecologic malignancy enrolled in surgical list of our institute
* must be able to consume oral supplements.

Exclusion Criteria:

* women that are not able to follow ERAS protocol due to medical reasons
* patients with severe disease that cannot compromise with protocol

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Perioperative infections | Postoperatively (30 days)
  We will notice possible surgical site infections,respiratory inflammations etc and calculate inflammatory markers and the concentration of white blood cells
Duration of hospitalization | Until discharge from hospital
  From date of hospitalization until the date of discharge or date of death from any cause, whichever came first, assessed up to 2 months.

SECONDARY OUTCOMES:
Postoperative mobilization | Until first day of mobilization
  From date of surgery until the date of discharge or date of death from any cause, whichever came first, assessed up to 2 months.
Postoperative morbidity (other than infectious) | 30 days
  Major events such as pulmonary embolism,accuse myocardial infarction,etc
Recurrence rates | 3 years follow-up
  Recurrent disease will be monitored through 3 year of follow up
Overall survival | 3 years follow-up
  Overall survival of the patients will be measured through 3 year of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Thomakos, Pf, Study Director — National Kapodistrian University of Athens,1st obs and gyn department
Locations (1):
- First department of Obstetrics and Gynecology, Athens, Greece

IPD SHARING:
Plan to Share IPD: No
Individual patient data will become available upon reasonable request

REFERENCES:
- [Background] Gupta R, Senagore A. Immunonutrition within enhanced recovery after surgery (ERAS): an unresolved matter. Perioper Med (Lond). 2017 Dec 11;6:24. doi: 10.1186/s13741-017-0080-5. eCollection 2017. PMID 29238571
- [Background] Moya P, Soriano-Irigaray L, Ramirez JM, Garcea A, Blasco O, Blanco FJ, Brugiotti C, Miranda E, Arroyo A. Perioperative Standard Oral Nutrition Supplements Versus Immunonutrition in Patients Undergoing Colorectal Resection in an Enhanced Recovery (ERAS) Protocol: A Multicenter Randomized Clinical Trial (SONVI Study). Medicine (Baltimore). 2016 May;95(21):e3704. doi: 10.1097/MD.0000000000003704. PMID 27227930
- [Background] Yeung SE, Hilkewich L, Gillis C, Heine JA, Fenton TR. Protein intakes are associated with reduced length of stay: a comparison between Enhanced Recovery After Surgery (ERAS) and conventional care after elective colorectal surgery. Am J Clin Nutr. 2017 Jul;106(1):44-51. doi: 10.3945/ajcn.116.148619. Epub 2017 May 3. PMID 28468890
- [Background] Fiorindi C, Cuffaro F, Piemonte G, Cricchio M, Addasi R, Dragoni G, Scaringi S, Nannoni A, Ficari F, Giudici F. Effect of long-lasting nutritional prehabilitation on postoperative outcome in elective surgery for IBD. Clin Nutr. 2021 Mar;40(3):928-935. doi: 10.1016/j.clnu.2020.06.020. Epub 2020 Jul 1. PMID 32684485
- [Background] Nelson G, Bakkum-Gamez J, Kalogera E, Glaser G, Altman A, Meyer LA, Taylor JS, Iniesta M, Lasala J, Mena G, Scott M, Gillis C, Elias K, Wijk L, Huang J, Nygren J, Ljungqvist O, Ramirez PT, Dowdy SC. Guidelines for perioperative care in gynecologic/oncology: Enhanced Recovery After Surgery (ERAS) Society recommendations-2019 update. Int J Gynecol Cancer. 2019 May;29(4):651-668. doi: 10.1136/ijgc-2019-000356. Epub 2019 Mar 15. PMID 30877144
- [Background] Nelson G, Fotopoulou C, Taylor J, Glaser G, Bakkum-Gamez J, Meyer LA, Stone R, Mena G, Elias KM, Altman AD, Bisch SP, Ramirez PT, Dowdy SC. Enhanced recovery after surgery (ERAS(R)) society guidelines for gynecologic oncology: Addressing implementation challenges - 2023 update. Gynecol Oncol. 2023 Jun;173:58-67. doi: 10.1016/j.ygyno.2023.04.009. Epub 2023 Apr 21. PMID 37086524